CLINICAL TRIAL: NCT06864858
Title: Clinical Evaluation of Two Cosmetic Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6571
Record Dates: First submitted 2025-02-14; First posted 2025-03-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Test Lens/Control Lens (Experimental): Eligible subjects will be randomized into the Test Lens/Control Lens sequence, to wear the Test Lens followed by the Control Lens in a bilateral fashion, with a washout period of 5-minutes between wear periods.
  Interventions: Device: etafilcon A with PVP with cosmetic pattern contact lens; Device: 1-DAY ACUVUE® DEFINE® with LACREON®, FRESH Honey
- Control Lens/Test Lens (Experimental): Eligible subjects will be randomized into the Control Lens/Test Lens sequence, to wear the Control Lens followed by the Test Lens in a bilateral fashion, with a washout period of 5-minutes between wear periods.
  Interventions: Device: etafilcon A with PVP with cosmetic pattern contact lens; Device: 1-DAY ACUVUE® DEFINE® with LACREON®, FRESH Honey

INTERVENTIONS:
Device: etafilcon A with PVP with cosmetic pattern contact lens — Test Lens
Device: 1-DAY ACUVUE® DEFINE® with LACREON®, FRESH Honey — Control Lens

SUMMARY:
This is a single visit, single-masked, non-dispensing, randomized, controlled, 2×2 bilateral crossover study to evaluate visual acuity.

ELIGIBILITY:
Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 39 (inclusive) years of age at the time of screening.
4. Be a current soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week over the last 30 days by self-report.
5. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 D to -6.00 D (inclusive) in each eye.
6. The subject's refractive cylinder must be less than or equal to 0.75 D (inclusive) in each eye.
7. Have spherical best corrected visual acuity of 20/25 or better in each eye.

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or lactating.
2. Have any systemic disease (eg, Sjögren's Syndrome), allergies, infectious disease (eg, hepatitis, tuberculosis), contagious immunosuppressive diseases (eg, HIV), autoimmune disease (eg rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study (at the investigator's discretion).
3. Use of systemic medications (eg, chronic steroid use) that are known to interfere with contact lens wear (at the investigator's discretion).
4. Have any previous, or planned (during the study), ocular surgery (eg, radial keratotomy, PRK, LASIK, etc.).
5. Have any previous history or signs of a contact lens-related corneal inflammatory event (eg, past peripheral ulcer or round peripheral scar), or any other ocular abnormality that would contraindicate contact lens wear (at the investigator's discretion).
6. Have participated in any contact lens or lens care product clinical trial within seven (7) days prior to study enrollment.
7. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
8. Have any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion (at the investigator's discretion).
9. Have any clinically significant (Grade 3 or 4 on FDA scale) tarsal abnormalities, bulbar injection, corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2025-03-30 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Visual Acuity (logMAR) | After approximately 90-minute lens wear period
  Monocular distance (4m) monocular VA under high-luminance high contrast (HLHC) will be measured post-lens fitting using ETDRS Charts.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- Maitland Vision Center - North Orlando Ave, Maitland, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu